CLINICAL TRIAL: NCT02633540
Title: A Phase II Investigation of Contralateral Arytenoid Sparing IMRT for T1a and T2a Larynx Cancer With Detailed Analysis of Post-treatment Laryngeal Function
Brief Title: Investigation of Contralateral Arytenoid Sparing IMRT for T1a & T2a Larynx Cancer & Analysis of Post-treatment Laryngeal Function
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-083; 15-1014 (Other: Fox Chase Cancer Center IRB)
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Laryngeal Neoplasms
Keywords: T1a Larynx Cancer; T2a Larynx Cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT Radiation (Experimental): All subjects will be treated using IMRT with the standard fractionation for T1a glottic cancer at Fox Chase Cancer Center: 63 Gy in 28 fractions; 6 for T1a and 65.25 Gy in 29 fractions; 33 for T2a. Treatment will be followed by functional assessments performed at months 1,3,6,12,and 24.
  Interventions: Radiation: IMRT Radiation

INTERVENTIONS:
Radiation: IMRT Radiation — Radiation to Larynx

SUMMARY:
The aim of this study is to define a new treatment technique for T1a larynx cancer that maintains excellent local control with less extensive radiation fields. It is thought that this will lead to patients having fewer changes to their voice and a higher quality of life after treatment when compared to the current standard treatment.

DETAILED DESCRIPTION:
Parallel opposed portal external beam radiation is the standard nonsurgical treatment for T1-2N0 glottic cancer. This technique involves treatment of the entire larynx for tumors that are small and limited. Although technological advances now allow radiation oncologists selectively to target and avoid adjacent sub-portions of any organ, these tools have not been applied T1-2N0 glottic cancer due to the perceived low toxicity of standard therapy. However, radiotherapy for early glottic cancer is not without functional side effects and it is not known whether post-treatment function after whole larynx radiation is superior to a more targeted surgical approach.

This is a phase II study to treat unilateral glottic cancer (Stage T1a and T2aN0) with intensity modulated radiation therapy (IMRT). In view of the anticipated small volume of disease at presentation and need to limit the potential for a "marginal miss", treatment will include the entire involved vocal fold, anterior commissure, and the anterior 1/3 of the contralateral vocal fold thus sparing the contralateral arytenoid cartilage and musculature ("contralateral arytenoid sparing IMRT"). In addition, we propose to perform sophisticated objective and patient reported measures regarding speech outcomes for two years after the completion of therapy at specified intervals, to better gain an understanding of the effects of therapy. Our findings will have the potential to dramatically advance the field of early larynx cancer therapy by demonstrating the efficacy of limiting the volume of uninvolved larynx that receives radiation and comprehensively assessing the functional outcomes of said therapy.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients with T1a or T2a squamous cell carcinoma of the glottic larynx (tumor limited to one vocal cord with normal cord mobility).
  * Patients must be able to read and write English to comply with the questionnaire portions of the protocol.
  * ECOG performance status of 0 or 1.
* Exclusion Criteria:

  * Patients with verrucous or adenocarcinoma
  * Patients with T1 tumors on both cords (T1b)
  * Patients with T2b-T4 true larynx tumors
  * Patients with primary supraglottic tumors that involve the true larynx
  * Patients with a prior or concurrent malignancy (other than nonmelanoma skin cancer or carcinoma in-situ of the cervix) are ineligible unless the previous cancer was treated 5 years or more prior to the current tumor and the patient has remained continually disease free
  * Patients who have received prior radiation to the head and neck
  * Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Galloway, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMRT Radiation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMRT Radiation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 48.5 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Voice Quality (Voice Handicap Index)
Description: Demonstrate a 50% improvement in the VHI (voice handicap index) score at 24 months after the completion of therapy IMRT for T1a/T2a larynx cancer
Time Frame: 24 Months
Population: Number of patients enrolled is too small for meaningful analysis
Arm/Group | IMRT Radiation
Number analyzed (Participants) | 0

2. Secondary Outcome: Patient-reported Swallowing Satisfaction
Description: Evaluate patient-reported satisfaction with swallowing at up to 24 months after the completion of radiation using the Eating Assessment Tool (EAT-10) questionnaire.
Time Frame: 24 Months
Population: Number of patients enrolled is too small for meaningful analysis
Arm/Group | IMRT Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinician Evaluation of Swallowing Function
Description: Evaluate clinician-reported measure of swallowing 24 months after the completion of radiation as measured by fiberoptic endoscopic evaluation of swallowing (FEES) using the penetration, aspiration scale (PAS) scores for 3 commonly evaluated textures (cookie, puree, thin).
Time Frame: 24 Months
Population: Number of patients enrolled is too small for meaningful analysis
Arm/Group | IMRT Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | IMRT Radiation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT02633540/Prot_SAP_000.pdf